CLINICAL TRIAL: NCT03851198
Title: Early Diagnosis of Patients With Mild Cognitive Impairment Through the Parameterization of Functional Tests.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants
Sponsor: University of Malaga (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IJFA07
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2020-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Diagnosis; Functional tests; Kinematics; Validation; Reliability
MeSH Terms: conditions — Cognitive Dysfunction; Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Cognitive Impairment patients (Experimental): Subjects diagnosed with mild cognitive impairment, who will receive the best treatment of clinical practice, will be recruited. They must be more than 60 years old.
  Interventions: Procedure: Standard Care or Usual Clinical Practice
- Healthy Subjects/ Match control (Active Comparator): Healthy subjects of the same age as people with mild cognitive impairment.
  Interventions: Procedure: Standard Care or Usual Clinical Practice

INTERVENTIONS:
Procedure: Standard Care or Usual Clinical Practice — The guidelines for the management according to the mild cognitive impairment in primary care will be the treatment guidelines for the Standard Care.

SUMMARY:
The present study aims to develop an index formed by the variables, functional tests, scales and instruments that best discriminate between healthy subjects and subjects with MCI and that allows the stratification of different levels of severity of MCI, and to validate new systems for the early diagnosis of subjects with mild cognitive impairment.

DETAILED DESCRIPTION:
Dementia affects 46.8 million people and in 2050 it is expected that there will be between 115-135 million people suffering from dementia. Inside dementias, Mild Cognitive Impairment (MCI) has a prevalence in adults aged ≥65 years of 10-20%.

Patients with MCI also show greater progression towards dementia, higher mortality and disability, and a greater use of medical care compared to cognitively normal subjects that converts MCI into an important public health problem, which reinforces the need to perfect clinic assessment procedures to improve the early identification of individuals with MCI. Early diagnosis could allow effective medical treatments that prevent or slow the onset of dementia, and could improve the effectiveness of non-pharmacological interventions.

Currently, it can be used an Inertial Sensor and 3D motion capture systems with a camera to analyse kinematics and these instruments are being integrated as a rehabilitation tool in patients. The use of Inertial Sensor and 3D motion capture cameras would help to find fast and cheap assessment methods for professionals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 60 years of age.
* Healthy subjects and subjects diagnosed with mild cognitive impairment.
* Subjects able of filling out questionnaires and performing functional tests.

Exclusion Criteria:

* Participants with neurological pathologies other than mild cognitive impairment.
* Participation in an experimental study where they receive a treatment.
* Score on the Mini-Mental State Examination of less than 24.
* Inability to get up from the chair at least 5 times or 30 seconds
* Inability to walk 20 meters.
* Inability to raise up both arms to 90 degrees or lifting 2 kg with the hand.
* Inability to walk independently without a walking assistance device (cane, crutch or walker).
* Patients with prescription of beta-blockers.
* Inability to provide informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Kinematic analysis by motion sensor | 1 hour
  An Inertial Sensor will pick up positioning, motion and acceleration information from the subject
Kinematic analysis by 3D motion capture | 1 hour
  The camera will perform a motion capture of the functional task. This system will calculate the displacement and the time of the functional task.
Responsiveness | 1 hour
  The Responsiveness Box of COSMIN checklist will be used to determinate the response to change of the Inertial Sensor and the 3D cameras. All possible items will be followed.
Reliability | 1 hour
  The Reliability Box of COSMIN checklist will be used to determinate the Test-Retest reliability of the Inertial Sensor and the 3D cameras. All possible items will be followed.
Validity | 1 hour
  The Criterion Validity Box of COSMIN checklist will be used to determinate the correlation between data from the Inertial Sensor and the 3D camera. All possible items will be followed.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 15 min
  Questionnaire used for the cognitive state assessment. The Mini-Mental State Examination includes eleven questions. The maximum total score is 30 points. It is divided into two sections, the first of which requires only vocal responses and covers orientation, memory and attention; the maximum score is 21. The second part assess the ability to name, follow verbal and written commands, write a sentence spontaneously and copy a complex polygon similar to a Bender-Gestalt figure; the maximum score is 9. As usual, a score lower 24 points points is indicatives of dementia.
Geriatric Depression Screening Scale (GDSS) | 15 min
  A questionnaire designed to detect depression in older adults. This scale consists of 30 items (answer format yes / no). Less score is indicative of depression. Generally, a score below 15 points is already indicatives of depression.
Katz Index | 15 min
  It is a hetero-administered questionnaire used to assess activities of daily living that includes 6 dichotomous items (bathing, dressing, goimt to toilet, transfer, continence, feeding). It is scored considering the items individually, so that 0 points are given when the activity is performed independently and 1 point if the activity is done with help or not done. The score varies from 0 to 6 points, with a higher score indicative of greater dependence on the development of activities of daily living.
Lawnton & Brody Scale | 15 min
  It is a hetero-administered questionnaire used to assess instrumented activities of daily living that includes the assessment of 8 activities of daily living (ability to use the telephone, shopping, food preparation, housekeeping, laundry, mode of transporation, responsibility for own medications and ability to handle finances). The score varies from 0 to 8 points. 0 points are given when the activity is performed independently and 1 point if the activity is done with help or not done. There is no cut-off point, but a higher score is indicative of worse performance of instrumental activities or less functionality.
Cardiopulmonary function | 1 hour
  The heart rate will be assessed using the Polar wrist heart rate monitor
Metabolic parameters | 1 hour
  The blood lactate produced will be analysed using the Lactate Pro 2 blood lactate analyzer
Sonographic parameters | 1 hour
  The thickness of the subcutaneous fat and the anterior rectus quadriceps muscle, and the eco-intensity of the subcutaneous fat and the anterior rectus quadriceps muscle, both at rest and in maximum voluntary isometric contraction, will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science School , University of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the anonymised data that conform the results that will be analysed in the present clinical trial, after the de-identification, will be published in a peer review journal (tables, figures, appendices, text). Moreover, data will be available to researchers who provide a methodologically sound proposal, but data will be not publicly available. Proposals will be directed by acuesta@uma.es. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months following article publication in a peer review jorunal. No definite end date.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. Proposals will be directed by acuesta@uma.es. To gain access, data requestors will need to sign a data access agreement.